CLINICAL TRIAL: NCT01002196
Title: How to Help When Silence is Not Golden A RCT Study of Selective Mutism
Brief Title: Randomised Controlled Treatment Study of Selective Mutism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regionsenter for barn og unges psykiske helse (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Hanne Kristensen, Director Section for Clinical Research, Regionsenter for barn og unges psykiske helse
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RegionsenterBUP; 190648/V50; Norwegian Research Council
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Selective Mutism
Keywords: Selective Mutism; Intervention
MeSH Terms: conditions — Mutism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- stimulus fading procedures (Experimental)
  Interventions: Behavioral: Stimulus fading procedures; Behavioral: Guidance on defocused communication
- guidance of defocused communication (Active Comparator)
  Interventions: Behavioral: Guidance on defocused communication

INTERVENTIONS:
Behavioral: Stimulus fading procedures — Core elements : 1.Behavior techniques (BT's) are used to gradually master the anxiety ("stimulus fading" and reward).
  2. Children are first met at home where they feel most safe, and the BT's are first conducted at home in cooperation with the parents.
  3.The same interventions are then continued in the environment where the problem primarily exist (kindergarten / school) not at the clinic.
  4.Defocused communication- and interaction is a general treatment principle (e.g. avoid looking directly at the child, sit beside not opposite to the child, no direct questioning, and communication is based upon a motivating activity, not about the child).
  5.Frequent and short interventions. 6.Information to parents and teachers on how to communicate with children with SM
  Other Names: stimulus fading technique; defocused communication
  Arms: stimulus fading procedures
Behavioral: Guidance on defocused communication — Guidance and supervision to teachers working with the children with SM. Frequency: Twice during three months

SUMMARY:
Selective mutism (SM) describes inhibited and withdrawn children who are persistently mute in central situations despite ability to talk. SM may cause great suffering and create problems, both socially and related to learning. SM is associated with social anxiety, neurodevelopmental delay and bilingualism. The prevalence is about .7-8 ‰. Adequate assessment and treatment of SM is seldom provided in the mental health services. SM is considered hard to treat, and randomised treatment studies are lacking. This study will examine the effect of a manual based treatment for SM. The treatment consists of home- and kindergarten /school based interventions including behaviour techniques and psychoeducation. Defocused communication is a general treatment principle. Comorbidity, including neurodevelopmental delay /disorder, and predictors of outcome, will be examined. A pilot study was conducted to ensure the feasibility of the planned effectiveness study. Seven children, aged 3-5 years were included. Six has started treatment, and all talked in the kinder garden within the first 3 months. The present study will have a randomised controlled design with 1. Manual based intervention for 6 months compared to 2. Waiting list controls (3 months), and then manual based intervention. The sample: Children aged 3-9 years consecutively referred to the school psychology- or the mental health services in Oslo and Eastern Norway. Expected N = 24 based on the pilot study, is a sufficient sample size to answer our primary research question. The treatment will be given by a therapist from the research group or by a local clinician under supervision. The study can add essential knowledge on treatment of SM and make effective treatment available to clinicians in the community.

ELIGIBILITY:
Inclusion Criteria:

* Children from Eastern & Southern Norway will be included if they fulfill the diagnostic criteria for SM

Exclusion Criteria:

* Children with SM and mental retardation with IQ below 50.
* Children with SM and psychosis or pervasive developmental disorders with the exception of Asperger syndrome and PDD Nos (DSM-IV)
* Children with SM who receive an active treatment for SM in the CAMHS
* Children with SM who are medicated for social anxiety.
* Children with SM where the parents do not understand Norwegian.

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
School version of the Selective Mutism Questionnaire (SSQ) | at 3, 6, 12 months

SECONDARY OUTCOMES:
Clinical Global Impression Scale (CGI) | at 3, 6, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Kristensen, MD, PhD, Principal Investigator — Regional Centre for Child and Adolescent Mental Health, Eastern and Southern Norway
Locations (1):
- Centre for Child and Adolescent Mental Health, Eastern and Southern Norway, Oslo, Norway

REFERENCES:
- [Derived] Oerbeck B, Stein MB, Wentzel-Larsen T, Langsrud O, Kristensen H. A randomized controlled trial of a home and school-based intervention for selective mutism - defocused communication and behavioural techniques. Child Adolesc Ment Health. 2014 Sep;19(3):192-198. doi: 10.1111/camh.12045. Epub 2013 Oct 26. PMID 32878377
- [Derived] Oerbeck B, Overgaard KR, Stein MB, Pripp AH, Kristensen H. Treatment of selective mutism: a 5-year follow-up study. Eur Child Adolesc Psychiatry. 2018 Aug;27(8):997-1009. doi: 10.1007/s00787-018-1110-7. Epub 2018 Jan 22. PMID 29357099
- [Derived] Oerbeck B, Stein MB, Pripp AH, Kristensen H. Selective mutism: follow-up study 1 year after end of treatment. Eur Child Adolesc Psychiatry. 2015 Jul;24(7):757-66. doi: 10.1007/s00787-014-0620-1. Epub 2014 Sep 30. PMID 25267381